CLINICAL TRIAL: NCT06131866
Title: The Effect of Acceptance and Commitment Therapy Based Psychoeducation on Meaning and Purpose of Life and Coping Skills in Patients With Bipolar Disorder
Brief Title: Acceptance and Commitment Therapy Based Psychoeducation, Meaning of Life and Coping Skills in Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kubra TOHUMCU (Other)
Responsible Party: Sponsor-Investigator, Kubra TOHUMCU, Nurse, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GAÜN KThmc
Record Dates: First submitted 2023-11-03; First posted 2023-11-14 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Bipolar Disorder; Coping Skills
Keywords: Bipolar Disorder; Copin Skills; Meaning and Purpose of Life; Acceptance and Commitment Therapy; Psychoeducation; Randomised Controlled Trial
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial consisting of a total of 8 groups, 4 experimental and 4 control
Who Masked: Participant
Masking Description: A total of 8 groups, 4 intervention groups and 4 control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- intervention group 1 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): After explaining the purpose of the study to the individuals, after obtaining their consent, "Personal Information Form", "Coping Attitudes Evaluation Scale COPE-R" and '' The pre-test will be applied by applying the "Meaning and Purpose of Life Scale", then the 8-week Acceptance and Commitment Therapy Based Psychoeducation programme will be applied and the post-test data will be collected. In the 12th week, follow-up test will be applied and evaluation will be made.
  Interventions: Other: Psychoeducation based on Acceptance and Commitment Therapy
- Control group 1 (No Intervention): After explaining the purpose of the study to the individuals participating in the study, after obtaining their consent, "Personal Information Form", "Coping Attitudes Evaluation Scale COPE-R" and '' Meaning and Purpose of Life Scale'' will be applied and pre-tests will be applied. Then, the post-test will be applied 8 weeks later without any intervention. One month after the post-test, i.e. at the 12th week, a follow-up test will be applied and an evaluation is planned.
- Intervention group 2 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): After explaining the purpose of the study to the individuals, after obtaining their consent, "Personal Information Form", "Coping Attitudes Evaluation Scale COPE-R" and '' The pre-test will be applied by applying the "Meaning and Purpose of Life Scale", then the 8-week Acceptance and Commitment Therapy Based Psychoeducation programme will be applied and the post-test data will be collected. In the 12th week, follow-up test will be applied and evaluation will be made.
  Interventions: Other: Psychoeducation based on Acceptance and Commitment Therapy
- Control group 2 (No Intervention): After explaining the purpose of the study to the individuals participating in the study, after obtaining their consent, "Personal Information Form", "Coping Attitudes Evaluation Scale COPE-R" and '' Meaning and Purpose of Life Scale'' will be applied and pre-tests will be applied. Then, the post-test will be applied 8 weeks later without any intervention. One month after the post-test, i.e. at the 12th week, a follow-up test will be applied and an evaluation is planned.
- Intervention group 3 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): After explaining the purpose of the study to the individuals, after obtaining their consent, "Personal Information Form", "Coping Attitudes Evaluation Scale COPE-R" and '' The pre-test will be applied by applying the "Meaning and Purpose of Life Scale", then the 8-week Acceptance and Commitment Therapy Based Psychoeducation programme will be applied and the post-test data will be collected. In the 12th week, follow-up test will be applied and evaluation will be made.
  Interventions: Other: Psychoeducation based on Acceptance and Commitment Therapy
- Control group 3 (No Intervention): After explaining the purpose of the study to the individuals participating in the study, after obtaining their consent, "Personal Information Form", "Coping Attitudes Evaluation Scale COPE-R" and '' Meaning and Purpose of Life Scale'' will be applied and pre-tests will be applied. Then, the post-test will be applied 8 weeks later without any intervention. One month after the post-test, i.e. at the 12th week, a follow-up test will be applied and an evaluation is planned.
- Intervention group 4 in which psychoeducation based on acceptance and commitment therapy was applied (Experimental): After explaining the purpose of the study to the individuals, after obtaining their consent, "Personal Information Form", "Coping Attitudes Evaluation Scale COPE-R" and '' The pre-test will be applied by applying the "Meaning and Purpose of Life Scale", then the 8-week Acceptance and Commitment Therapy Based Psychoeducation programme will be applied and the post-test data will be collected. In the 12th week, follow-up test will be applied and evaluation will be made.
  Interventions: Other: Psychoeducation based on Acceptance and Commitment Therapy
- Control group 4 (No Intervention): After explaining the purpose of the study to the individuals participating in the study, after obtaining their consent, "Personal Information Form", "Coping Attitudes Evaluation Scale COPE-R" and '' Meaning and Purpose of Life Scale'' will be applied and pre-tests will be applied. Then, the post-test will be applied 8 weeks later without any intervention. One month after the post-test, i.e. at the 12th week, a follow-up test will be applied and an evaluation is planned.

INTERVENTIONS:
Other: Psychoeducation based on Acceptance and Commitment Therapy — Acceptance and Commitment Therapy Based Psychoeducation will be applied to the patients in the intervention group in the form of group education (consisting of 5-7 people), one session per week for eight weeks; no intervention will be applied to the control group.
  Arms: Intervention group 2 in which psychoeducation based on acceptance and commitment therapy was applied; Intervention group 3 in which psychoeducation based on acceptance and commitment therapy was applied; Intervention group 4 in which psychoeducation based on acceptance and commitment therapy was applied; intervention group 1 in which psychoeducation based on acceptance and commitment therapy was applied

SUMMARY:
This research will be conducted to determine the effect of acceptance and commitment therapy-based psychoeducation on coping skills and finding meaning in life in patients with bipolar disorder. This research is planned as a randomised controlled experimental study. The study will be conducted with euthymic stage patients diagnosed with bipolar disorder who applied to Adıyaman Besni State Hospital psychiatry outpatient clinic using randomisation method. According to the power analysis result, the study will be applied to a total of 40 individuals, 20 experimental and 20 control. "Individual Information Form" regarding socio-demographic characteristics, "Coping Attitudes Evaluation Scale COPE-R" and "Meaning and Purpose of Life Scale" will be used to collect the data. Acceptance and Commitment Therapy Based Psychoeducation will be applied to the patients in the intervention group in the form of group education (consisting of 5-7 people), one session per week for eight weeks; no intervention will be applied to the control group. Pre-tests will be applied to the patients in the intervention and control groups just before the training, post-test will be applied to the intervention group immediately after the training sessions are completed, and follow-up test will be applied one month after the post-test, i.e. in the 12th week. After the pre-test was applied to the control group, the post-test will be applied in the 8th week and the follow-up test will be applied in the 12th week without any intervention. In the evaluation of the data; descriptive statistical methods (frequency, mean), t-test, one way Anova and correlation analyses will be used. Permission was obtained from the University Ethics Committee, the relevant institution and the individuals participating in the study.

DETAILED DESCRIPTION:
Bipolar disorder negatively affects individuals' mental and physical health, interpersonal relationships, educational and occupational functions. Factors such as personality structure, coping with stress and social adaptation skills play an important role in the course of the disease as well as neurobiological factors. Bipolar disorder is a difficult condition for people to cope with due to its chronic nature and these individuals have problems in interpersonal relationships and coping with stress. Beyond what is perceived in relation to normal life, bipolar disorder causes individuals to experience large and complex extra dimensions in all aspects of their lives and to struggle for meaning in their lives. Three indicators of an individual's psychological well-being are the individual's goals in life, awareness of his/her existing potential and the quality of interpersonal relationships. In bipolar disorder, which also affects the psychological well-being of individuals, individuals often do not achieve complete remission despite pharmacotherapy. In addition to pharmacotherapy, various psychosocial interventions such as cognitive behavioural therapies and psychoeducation have been developed and applied to treat bipolar disorder. Acceptance and Commitment Therapy is one of the leading types of therapy methods called the third generation of cognitive behavioural therapies. Instead of teaching individuals to control their feelings, thoughts, sensations, memories and other subjective situations, acceptance and stability therapy teaches individuals to recognise and accept these experiences and, most importantly, to embrace their negative experiences. Acceptance and commitment therapy aims to change individuals' relationships with the emotions, thoughts, memories and physical sensations that they fear and avoid. It uses acceptance and awareness strategies to teach individuals to focus on the present moment and to reduce avoidance and cognitive attachment. Thus, individuals learn to clarify their goals and values and learn to adhere to behaviour change strategies. Acceptance and commitment therapy is one of the psychotherapies supported by the American Psychological Association for most psychiatric conditions, including psychosis. The transdiagnostic nature of acceptance and commitment therapy is compatible with mood disorders as well as psychotic symptoms. Acceptance and commitment therapy has been shown to be effective in many psychopathological conditions, including bipolar disorder. It is stated in the literature that an innovative group intervention combining acceptance and commitment therapy and psychoeducation approaches may be beneficial in individuals with bipolar disorder. Psychoeducational programmes are auxiliary interventions that complement pharmacological treatment in order to further reduce the burden of the disease and relapses in mental disorders. The effectiveness of psychoeducation in patients with bipolar disorder has been shown in many studies.

ELIGIBILITY:
Inclusion Criteria:

* To be receiving outpatient treatment with the diagnosis of Bipolar Disorder according to DSM-5
* Being in euthymic mood according to the doctor's control at the time of the interview
* Having no problem in understanding and speaking Turkish
* Being literate
* Being in the 18-65 age group
* Not having undergone such training for the last 1 year

Exclusion Criteria:

* Presence of serious sensory and cognitive disabilities that would prevent answering the questionnaire
* Refusal to participate in the study after being informed
* Having another psychiatric diagnosis in addition to the diagnosis of bipolar disorder
* Having an attack period during the education process

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
Acceptance and commitment therapy-based psychoeducation and the level of finding meaning in life in patients with bipolar disorder | up to 12 weeks
  The effect of acceptance and commitment therapy-based psychoeducation on individuals' levels of finding meaning in life in patients with bipolar disorder Personal Information Form and Meaning and Purpose of Life Scale pretests will be applied to the patients in the intervention group before the training. Afterwards, acceptance and stability-based psychoeducation consisting of 8 modules will be applied. Post-tests will be administered after the sessions and a follow-up test will be administered one month later (at the 12th week). Meaning and Purpose of Life Scale minimum score=17, maximum score=85. The high score obtained from the scale indicates that the level of meaning in the lives of individuals is high.

SECONDARY OUTCOMES:
Acceptance and commitment therapy-based psychoeducation and coping skills in patients with bipolar disorder | up to 12 weeks
  The effect of acceptance and commitment therapy-based psychoeducation on coping skills levels in patients with bipolar disorder Personal Information Form and Coping Attitudes Evaluation Scale COPE-R pretests will be applied to the patients in the intervention group before the training. Afterwards, acceptance and stability-based psychoeducation consisting of 8 modules will be applied. Post-tests will be administered after the sessions and a follow-up test will be administered one month later (at the 12th week). Coping Attitudes Rating Scale COPE-R minimum score=32, maximum score=128. The high score obtained from the scale indicates a high level of coping attitude.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No